CLINICAL TRIAL: NCT05698810
Title: Preparation and Feasibility of Exams for Expected Studies (PRELUDE)
Brief Title: Preparation and Feasibility of Exams for Expected Studies
Acronym: PRELUDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Commissariat A L'energie Atomique (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC22.0130
Record Dates: First submitted 2022-12-13; First posted 2023-01-26 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers; Parkinson's Disease Patients; Para/Tetraplegic Patients
MeSH Terms: interventions — Magnetoencephalography; Magnetic Resonance Spectroscopy; epicatechin gallate

STUDY DESIGN:
Intervention Model Description: volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Volunteers (Other): tests
  Interventions: Other: CE marked Medical Device MagnetoEncephaloGraphy (MEG) usability; Other: CE marked Medical Device Magnetic Resonance Imaging (MRI) usability; Other: CE marked Medical Device ElectroEncephaloGraphy (EEG) usability; Other: CE marked Medical Device ElectroCardioGraphy (ECG) usability
- Parkinson's Disease patients (Other): tests
  Interventions: Other: CE marked Medical Device MagnetoEncephaloGraphy (MEG) usability; Other: CE marked Medical Device Magnetic Resonance Imaging (MRI) usability; Other: CE marked Medical Device ElectroEncephaloGraphy (EEG) usability; Other: CE marked Medical Device ElectroCardioGraphy (ECG) usability
- Para/tetraplegic Patients (Other): tests
  Interventions: Other: CE marked Medical Device MagnetoEncephaloGraphy (MEG) usability; Other: CE marked Medical Device Magnetic Resonance Imaging (MRI) usability; Other: CE marked Medical Device ElectroEncephaloGraphy (EEG) usability; Other: CE marked Medical Device ElectroCardioGraphy (ECG) usability

INTERVENTIONS:
Other: CE marked Medical Device MagnetoEncephaloGraphy (MEG) usability — tests
Other: CE marked Medical Device Magnetic Resonance Imaging (MRI) usability — tests
Other: CE marked Medical Device ElectroEncephaloGraphy (EEG) usability — tests
Other: CE marked Medical Device ElectroCardioGraphy (ECG) usability — tests

SUMMARY:
Feasibility study: the examinations carried out as part of this protocol aim to carry out all the acquisitions and simulations of use, necessary for the development of the clinical research protocols to come to Clinatec (in particular, configuration of the equipment, dimension of the examination time and the size of the cohorts etc ...)

DETAILED DESCRIPTION:
To ensure the feasibility of a clinical trial, it is necessary to test the parameters as well as the sequence of the different examination times offered to participants.

The expected results of this protocol are mainly the dimension of experimental paradigms and the optimization of the clinical management of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ⩾ 18 years
* Affiliated to a social security scheme
* Free and informed consent signed

Exclusion Criteria:

* Subject in a period of exclusion from another study.
* Subject deprived of liberty by a judicial or administrative decision, or major subject subject to a legal protection measure (guardianship, curatorship and safeguarding of justice) referred to in Articles 1121-6 to 1121-8 of the Public Health Code.
* Subject who would receive more than 4500 euros in compensation because of his participation in other research involving the human person in the 12 months preceding this study.
* Pregnant woman, parturient, nursing mother (Article 1121-5 of the Public Health Code)
* Subject not reachable urgently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2033-03-20 (Estimated); Study Completion 2033-03-20 (Estimated)

PRIMARY OUTCOMES:
MEG physiological parameters measurements that will be used in future clinical research protocols | through study completion, an average of 10 years
  Adequacy of MEG physiological parameters measurements to the needs of the protocol and duration of the paradigm consistent with the cooperation of the subject
MRI physiological parameters measurements that will be used in future clinical research | through study completion, an average of 10 years
  Adequacy of MRI physiological parameters measurements to the needs of the protocol and duration of the paradigm consistent with the cooperation of the subject
EEG physiological parameters measurements that will be used in future clinical research | through study completion, an average of 10 years
  Adequacy of EEG physiological parameters measurements to the needs of the protocol and duration of the paradigm consistent with the cooperation of the subject
ECG physiological parameters measurements that will be used in future clinical research | through study completion, an average of 10 years
  Adequacy of ECG physiological parameters measurements to the needs of the protocol and duration of the paradigm consistent with the cooperation of the subject

SECONDARY OUTCOMES:
MEG physiological parameters data collection paradigms | through study completion, an average of 10 years
  Achieving MEG physiological parameters data collection paradigms
MRI physiological parameters data collection paradigms | through study completion, an average of 10 years
  Achieving MRI physiological parameters data collection paradigms
EEG physiological parameters data collection paradigms | through study completion, an average of 10 years
  Achieving EEG physiological parameters data collection paradigms
ECG physiological parameters data collection paradigms | through study completion, an average of 10 years
  Achieving ECG physiological parameters data collection paradigms

CONTACTS AND LOCATIONS:
Locations (1):
- Clinatec Cea/Chuga, Grenoble, France

IPD SHARING:
Plan to Share IPD: No